CLINICAL TRIAL: NCT00874913
Title: Study of Ocular Blood Flow Using Laser Doppler Flowmetry in Patients With Glaucoma and/or OSAS
Brief Title: Study of Ocular Blood Flow in Patients With Glaucoma and/or Obstructive Sleep Apnea Syndrome (OSAS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: DGS 2006/0052
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: blood flow; obstructive sleep apnea syndrome; normal tension glaucoma
MeSH Terms: conditions — Sleep Apnea, Obstructive; Low Tension Glaucoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser Doppler Flowmetry (Experimental)
  Interventions: Device: measurement of ocular blood flow

INTERVENTIONS:
Device: measurement of ocular blood flow — measurement of ocular blood flow with a laser Doppler flowmeter

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) is a common disease, with a prevalence evaluated between 5 - 7% in the general population. OSAS is characterized by recurrent episodes of partial or complete upper airway obstruction during sleep, which are nearly systematically associated with a desaturation-reoxygenation sequence, an admitted detrimental stimulus for the cardiovascular system. It has now been demonstrated that OSAS per se is able to generate hypertension, atherosclerosis and autonomic dysfunction (high sympathic tone and increase in baseline heart rate), all conditions possibly interacting with ocular vascular regulation. OSAS has major consequences on the ocular level since it is associated with a higher frequency of optic neuropathies, such as glaucoma and nonarteritic ischemic optic neuropathy (NAION), both with functional severe prognosis. Most of vascular changes associated with OSAS have been studied at the level of macrovasculature. In terms of physiopathology, the main effects on the vascular system in OSAS are sympathetic hyperactivity, oxidative stress, development of endothelial dysfunction, systemic inflammation and metabolic alterations such as the appearance of insulin resistance. All these mechanisms can affect the microcirculation of the eye, especially the optic nerve and choroid. Our hypothesis is that the eye microvasculature is affected by OSAS, and these lesions may be detected via a reduced autoregulation of blood flow in humans.

This project aims to demonstrate, quantify, and analyze the vascular modifications of the eye associated with OSAS trough a comparative clinical study on glaucoma patients and OSAS patients and matched healthy subjects for the regulation of the eye blood flow using confocal laser Doppler flowmetry (LDF). The regulation of the ocular blood flow will be assessed using several stimuli and measured using a new confocal LDF.

DETAILED DESCRIPTION:
JUSTIFICATION OF THE PROJECT Obstructive sleep apnea syndrome (OSA) is an under diagnosed disease affecting 5% of the general population. This disease is associated with an increase in the risk for cardiovascular disease (high blood pressure, coronary disease, and stroke). Two optic neuropathies are associated with OSA: glaucoma and nonarteritic anterior ischemic optic neuropathy (NAION). Glaucoma is a frequent progressive optical neuropathy in industrialized countries and one of the leading causes of blindness in the world. Normal tension glaucoma, a vascular form of glaucoma, is the form most frequently associated with OSAS. In addition, in nonglaucomatous OSA patients, there is a diffuse reduction in optic nerve layer thickness correlated with OSA severity, strongly suggesting optic nerve involvement in these patients. Moreover, recent studies have shown that 90% of patients presenting NAION have OSA. These clinical and epidemiological data suggest a causal relation between OSA and the onset of optic neuropathy.

OBJECTIVES: This physiopathological study aims to demonstrate, quantify, and analyze the vascular modifications associated with OSA through:

- A comparative study on glaucoma patients and OSAS patients, with or without NAION, and healthy subjects matched for age, sex, and body mass index: the eye vascular modifications will be quantified using confocal laser Doppler flowmetry.

EXPERIMENTAL SCHEDULE The aim of this study is to characterize ocular blood flow (choroid and optic nerve) regulation in patients in 4 populations: (1) glaucoma patients (2) OSA patients without clinical evidence of optic nerve disease, (3) OSA patients with NAION, (4) matched healthy subjects . OSA patients of group 2 and 3 will be studied 3-6 months after nCPAP treatment.

1. Recruitment and screening visit: each subject will undergo a general examination. The ocular examination includes visual acuity, intraocular pressure, biomicroscopy and fundus examination, visual field (Humphrey 24/2 SITA-STANDARD) and measurement of the thickness of the optic nerve fiber layer using optical coherence tomography (OCT 3 Zeiss). In order to assess the cardiovascular phenotype, the cardiovascular examination will be completed, by an electrocardiogram, an ambulatory blood pressure monitoring, and echocardiography. A blood sample will be also analyzed: lipid analysis, hemogram, ionogram, glucose, cholesterol, triglycerides. A polysomnography will be performed for all subjects for the diagnosis of OSA, and the calculation of a respiratory disturbance index (RDI, sleep apnea defined as a RDI >15 per hour).
2. Baseline measurements of blood flow of the optic nerve head:

   Patients are asked to abstain from alcohol and caffeine for at least 12 h before the LDF measurements. Systolic (BPsyst) and diastolic (BPdiast) blood pressures are determined (DINAMAP®, Critikon, inc. Tampa, Florida, USA) during LDF measurements and immediately after, intraocular pressure (IOP) of the fellow eye is measured by applanation tonometry: using the Tonopen XL. The mean ocular perfusion pressure (OPP) is calculated according to the formula: OPP sitting position = (95/140 x MAP) - IOP in which mean arterial pressure (MAP) was calculated as: MAP = BPdiast + 1/3 (BPsyst - BPdiast).

   A newly developed compact laser Doppler flowmeter (LDF) allows the measurement of blood flow at the level of the neuroretinal rim of the optic nerve. This system delivers a laser beam from a diode laser (670 nm) to a discrete site at the optic nerve head. The scattered light is collected by an optical fiber with the image of its aperture (approximately 150 µm in diameter) focused onto the illuminated site. This fiber guides the scattered light to a photodetector. An area of the fundus (30° in diameter) is illuminated in red-free light for observation of the fundus and positioning of the laser beam. This instrument detects the light scattered by the red blood cells (RBCs) within an annulus centered on the illumination site of the laser. This flowmeter consists of a self-aligned confocal system, a fundus illumination (green light) and CCD based observation unit, a target fixation system and a CCD camera to observe the pupil. This CCD allows monitoring of the position of the probing laser beam at the pupil to insure constant entrance point in successive measurements of ONH blood flow. The Doppler signal is digitized and a dedicated software operating on a portable computer calculates the relative velocity (VEL), volume (VOL) and flow of the red blood cells in the eye microcirculation. Synchronization of these parameters with the heart pulse allows determination of the flow pulsatility. For the investigation of the effect of increased retinal activity on optic nerve blood flow, a system for delivering visual stimuli (flicker) has been adapted to the fundus camera-based instrument.

   The baseline measurements consist on 3 measurements of the optic nerve blood flow in a resting condition every one minute during 3 minutes (time of measurement 30 sec).
3. Ocular blood flow reactivity: gas inhalation, isometric exercise and flicker stimulation.

   All these experiments will be performed in the 4 groups (glaucoma patients,OSA patients, patients with OSA+NAION, healthy subjects). A resting period of at least 20 minutes in a sitting position is scheduled for each subject before the study and 30 minutes between experiment. Stable baseline conditions are established, which are ensured by repeated measurements of blood pressure. Other conditions such as abstinence from coffee, alcohol drinking, smoking, refrain from heavy meal, exercise, etc, all of which may affect the measurement of blood flow are prohibited. Adequate dilatation of the patient's pupil is necessary using a muscarinic antagonist (i.e. tropicamide).

   The gas experiment

   - experimental setting : this experiment will be performed in a randomized, double masked, three way cross-over design. Three inhalation periods of different mixtures of oxygen and carbon dioxide are scheduled. Three LDF measurements of 30 seconds are performed before inhalation, 5 and 10 minutes during the inhalation, and then after resting period of 10 minutes. The following gas mixtures are administered for 10 minutes each: 100% O2, Bactal (92%O2 +8%CO2), and air (21,8%O2 +78,2%N2). All gases are delivered through a partially expanded reservoir bag at atmospheric pressure using a two valves system to prevent re-breathing. Transcutaneous carbon dioxide tension (TINA PtcCO2 monitoring system, Radiometer, Copenhagen, Denmark), MAP and IOP are monitored at 5', 10' and at the end of the experiment.

   The isometric exercise (handgripping)

   - experimental setting: this consists on handgripping during 3 minutes. Measurements of blood flow is performed each minute during a 30 sec period.

   The flicker experiment

   - experimental setting: The stimulus is a pure green luminance flicker generated by an array of ultrabright light-emitting diodes with dominant wavelengths at 524 nm and located in the plane of the light source of the fundus camera. The diodes are synchronously square-wave modulated at 15 Hz between 0 and 10 lux. The stimulus is delivered to the eye in Maxwellian view through the fundus illumination's optical system of the camera (Topcon Optical, Tokyo, Japan) and it uniformly illuminates a 25° diameter area that included both the fovea and the optic disc. Blood flow is measured at baseline before the flicker stimulation, and then during the 2 min period of flicker stimulation.
4. Similar experiments will be also performed for the OSA group of patients after 3 to 6 months of nCPAP treatment.

STUDIED POPULATION :

This clinical project will include OSA patients with the following inclusion criteria: OSA defined by a respiratory-disturbance index > 15/hour (number of episode of partial (hypopnea) or complete (apnea) upper airway obstruction), age between 18 and 80 years, affiliation to the health care system. The exclusion criteria are: ocular disease (including cataract or retinal disease, ametropia > 3 diopters, optic neuropathy other than NAION in group 2), uncontrolled high blood pressure, cardiovascular treatment (vasoconstrictors, vasodilatators, beta and alpha agonists or antagonists, nitric derived medication), corticosteroids, theophylline, sildenafil, immunosuppressors, neuroleptics, non steroid anti inflammatory, oestroprogestative treatment, hypnotics (benzodiazepines), local treatment for ocular hypertension or glaucoma.

Glaucoma was defined as:

Patients were eligible if they had glaucomatous optic nerve head appearance indicative of glaucoma in addition to corresponding visual field loss.

Visual field abnormalitie(s) compatible with glaucomatous damages in accordance to the European guidelines :

Unless one of the following criteria, observed on 2 consecutive automated visual fields (one of these will be the baseline automated visual field: Humphrey 30.2 SITA-Standard strategy):

* A Glaucoma Hemifield Test (GHT) outside normal limits. or
* A cluster of 3 or more nonedge points in a location typical for glaucoma, all of which are depressed on the pattern deviation plot at a p < 5% level and 1 of which is depressed at a p < 1% level.

or

- A Pattern Standard Deviation (PSD) that occurs in less than 5% of normal fields

Control subjects will be matched with OSA patients for body mass index, gender and age, and will undergo complete overnight polysomnography to discard OSA. Other inclusion and exclusion criteria are similar to that of OSA patients.

MAIN CRITERIA OF EVALUATION AND STATISTICAL ANALYSIS Normalized data during the experiment will be calculated according to baseline data. Changes in blood flow parameters (reflected the vascular reactivity) and correlations will be calculated with nonparametric tests (Friedman and Wilcoxon tests for paired comparisons) using the SPSS 12.0 software. Comparison of OSA group and healthy subjects group will be done using non parametric test (Mann Whitney and Chi 2 test). A two-tailed approach test will determine significance, which is set as p<0.05.

The sensitivity (the minimum statistically significant LDF parameters change (S) that can be detected) will be calculated using the formula : S = (t * SD) / ((square root)n * P mean) * 100, where P mean is the mean value of all measurements, SD the SD of the difference between paired measurement for all subjects, and t the two-tailed value of the t distribution at a 0.05 significance level for n-1-1 degree of freedom.

STRATEGY OF ANALYSIS The clinical experiment aims to compare the vascular regulation of the optic nerve in OSA patients with that of a healthy group of human subjects. Subsequently, a group of OSA patients with NAION will be analyzed in order to compare the ocular blood flow ant its regulation in eyes with ischemic neuropathy (NAION) with eyes of OSA patients without optic nerve disease. All these comparisons will allow to characterize the optic nerve blood flow in healthy eyes, in eyes of OSA patients and in eyes of OSA patients at the time of acute ischemic attack (NAION).The glaucoma patients will be compared with healthy subjects.

ETHICAL ASPECTS This study will be conducted in accordance with the Declaration of Helsinki for research involving human subjects and the Good Clinical Practice guidelines. Informed consent will be obtained from the subjects after explanation of the study. The study protocol was approved by the local Institutional Review Board (Comité de Protection des Personnes, Sud-Est V), declared to the French authorities (insurance : N° contract : 124706 Société Hospitalière d'Assurances Mutuelles Lyon, France).

ELIGIBILITY:
Inclusion Criteria:

1. the age is between 18 years & 80 years
2. nobody affiliated with social security
3. including informed & signed consent

Exclusion Criteria:

1. congenital malformation leading to an excavation of the optic nerve or a deficit of the visual field
2. any eye disease associated, including refraction disorder ( > 4 diopters) , retinal disease, cataract, corneal opacity)
3. taking medication which can have an action on blood pressure or regulation ( vasoconstrictors, vasodilators, beta-agonists and antagonists, nitrates, theophylline, dipyridamole, sildenafil, immunosuppressive, corticosteroid or Non-steroidal anti-inflammatory drugs (> 10 days), hormonal therapy), sedative drug (antidepressive, anxiolytics, hypnotics) drops with activity on regulation of ocular pressure ( beta-blockers)
4. all ophthalmic drops
5. pregnancy
6. current infection ( acute hepatitis B, hepatitis C active, HIV infection)
7. known hypertension or suspected
8. Electrolyte disturbance
9. Pathology that can affect the regulation of blood pressure : parkinson' disease, patients transplanted kidney or cardiac arrhythmias, severe heart failure atrial fibrillation or frequent extrasystole (> 10 / minute)
10. nocturnal Professional activity
11. History of surgery or carotid stenting
12. Previous treatment of Obstructive Sleep Apnea Syndrome by continuous positive pressure, propulsion prosthesis mandibular or maxillofacial surgery
13. No predictable compliance with the protocol
14. Patients participating in another biomedical research
15. Patients with no affiliation to social security
16. narrow irido corneal angle

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-09; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
ocular blood flow | 9 months

SECONDARY OUTCOMES:
comparisons between OSAS patients and healthy controls | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Romanet, Professor, MD, Principal Investigator — ophthalmology service, university hospital, grenoble; Christophe CHIQUET, Professor, MD, PhD, Study Chair — Ophthalmology service, University hospital, Grenoble; Karine Palombi, Doctor, MD, Principal Investigator — ophthalmology service, university hospital, grenoble; Elisabeth Renard, Doctor, MD, Principal Investigator — ophthalmology service, university hospital, grenoble; Jean-Louis Pepin, Professor, MD, PhD, Study Director — sleep laboratory, university hospital, grenoble; Patrick Levy, Professor, MD, PhD, Principal Investigator — sleep laboratory, university hospital, grenoble; Renaud Tamisier, Doctor, MD, PhD, Principal Investigator — sleep laboratory, university hospital, grenoble; Jean-Philippe Baguet, Professor, MD, PhD, Principal Investigator — cardiology service, university hospital, grenoble
Locations (1):
- Chu de Grenoble, Grenoble, France

REFERENCES:
- [Derived] Chiquet C, Lacharme T, Riva C, Almanjoumi A, Aptel F, Khayi H, Arnol N, Romanet JP, Geiser M. Continuous response of optic nerve head blood flow to increase of arterial blood pressure in humans. Invest Ophthalmol Vis Sci. 2014 Jan 23;55(1):485-91. doi: 10.1167/iovs.13-12975. PMID 24355824
- [Derived] Khayi H, Pepin JL, Geiser MH, Tonini M, Tamisier R, Renard E, Baguet JP, Levy P, Romanet JP, Chiquet C. Choroidal blood flow regulation after posture change or isometric exercise in men with obstructive sleep apnea syndrome. Invest Ophthalmol Vis Sci. 2011 Dec 16;52(13):9489-96. doi: 10.1167/iovs.11-7936. PMID 22025580